CLINICAL TRIAL: NCT02503904
Title: Tumescent Antibiotic Delivery for Prevention of Surgical Site Infection: A Multicenter Open Label Randomized Clinical Trial
Brief Title: Tumescent Antibiotic Delivery for Prevention of Surgical Site Infection
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Klein, Jeffrey A., M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TAD4SSI
Record Dates: First submitted 2014-12-26; First posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Surgical Site Infections; Venous Thromboembolism
Keywords: Pharmacology; Lidocaine; Epinephrine; Cefazolin; Metronidazole; Infection; prevention; prophylaxis; SSI; Surgery; Complications
MeSH Terms: conditions — Surgical Wound Infection; Venous Thromboembolism; Infections | interventions — Parturition; Metronidazole; Epinephrine; Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAD+IVAD (Active Comparator)
  Interventions: Procedure: Concomitant Tumescent Antibiotic Delivery & IV Delivery; Device: Subcutaneous Tumescent Infiltration; Drug: cecefazolin and metronidazole (in a dilute solution of tumescent lidocaine, epinephrin and sodium bicarbonate in 0.9% physiologic saline)
- IVAD (Active Comparator)
  Interventions: Procedure: Concomitant Tumescent Antibiotic Delivery & IV Delivery; Drug: cecefazolin and metronidazole (in a dilute solution of tumescent lidocaine, epinephrin and sodium bicarbonate in 0.9% physiologic saline)

INTERVENTIONS:
Procedure: Concomitant Tumescent Antibiotic Delivery & IV Delivery — Concomitant subcutaneous infiltration of a dilute antibiotics (cefazolin and metronidazole) in a dilute solution of tumescent lidocaine and epinephrine at the site of a proposed surgical incision.
  Other Names: TAD+IVAD
Device: Subcutaneous Tumescent Infiltration — Subcutaneous tumescent infiltration using HK tumescent infiltration cannulas and HK tumescent infiltration pump
  Arms: TAD+IVAD
Drug: cecefazolin and metronidazole (in a dilute solution of tumescent lidocaine, epinephrin and sodium bicarbonate in 0.9% physiologic saline)

SUMMARY:
The principal aim of the present research is to compare two methods of antibiotic delivery: concomitant tumescent antibiotic delivery (TAD) and intravenous antibiotic delivery (IVAD) versus IVAD alone, (TAD+IVAD vs IVAD), with respect to the prevention of surgical site infections (SSI). The investigators hypothesize that TAD+IVAD will significantly reduce the incidence of SSI compared to IVAD.

TAD is the subcutaneous infiltration of a dilute solution of antibiotic(s) in a solution of tumescent local anesthesia (TLA). TLA consists of a dilute solution of lidocaine (1gm/L), epinephrine (1mg/L) and sodium bicarbonate (10mEq/L) in 0.9% physiologic saline.

A secondary aim of this study is to compare TAD+IVAD vs IVAD with respect to the prevention of post-operative venous thromboembolism (VTE).

DETAILED DESCRIPTION:
Tumescent antibiotic delivery (TAD) is defined as the subcutaneous infiltration of a dilute solution of antibiotic(s) in a solution of tumescent local anesthesia (TLA). TLA consists of a dilute solution of lidocaine (1gm/L), epinephrine (1mg/L) and sodium bicarbonate (10mEq/L) in 0.9% physiologic saline.

The investigators hypothesize that TAD with intravenous antibiotic delivery (IVAD) will significantly reduce the incidence of SSI.

The Principal aim of the present research is to compare two methods of antibiotic delivery: concomitant TAD and IVAD versus IVAD alone (TAD+IVAD vs IVAD) with respect to the prevention of surgical site infections (SSI). The secondary aim of this study is to compare TAD+IVAD vs IVAD with respect to the prevention of post-operative venous thromboembolism (VTE). This research is an open label randomized clinical trial (RCT) comparing two modes of antibiotic delivery. It is not a trial comparing antibiotics.

The target populations for the present clinical trial are patients who have a high risk of SSI. These include patients exposed to high-risk surgical procedures (open abdominal surgeries, trauma surgeries, burn surgeries, sternotomy) or are obese, have diabetes, are immune-compromised or are otherwise at increased risk of SSI.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects greater than 18 years of age scheduled for surgical procedure considered to have a high risk for a surgical site infection (SSI) such as 1) secondary repair of a ventral hernia, 2) open bariatric surgery, 3) open abdominal colorectal surgery, 4) trauma surgery, 5) burn surgery or 6) sternotomy.

  2. Patients must have one of the following risk factors for surgical site infection: emergency surgery, obesity, diabetes mellitus, cancer surgery, be immune-compromised or otherwise be at an increased risk for SSI.

  3. Only adults will participate as research subjects 4. This study will involve both males and females 5. Patients in ASA (American Society of Anesthesiology) class I or II or III or IV will be included. Treatment assignment will be stratified with respect to ASA classification.

  6. Abdominal wound classifications: Clean-Contaminated, Contaminated, or Dirty are eligible to participate. Treatment assignment will be stratified with respect wound classification. Similarly, trauma and burn patients will be classified.

  7. Patient must be able to understand the same written and spoken language as either the surgeon or nurse who provides informed-consent information to the patient.

  8. Patients must be appropriately screened for the proposed surgery.

Exclusion Criteria:

Procedures involving only simple ostomy closures 2. Known allergy to cefazolin or metronidazole or an antibiotic preferred and routinely used by the surgeon 3. Persons less than 18 years old 4. Emergency operation as designated by the surgeon will be included only with the appropriate approval by the institutional IRB at an individual research site 5. Pregnant or breast-feeding women 6. A known bleeding/hemorrhagic/thrombotic disorder is exclusionary unless there is a written clearance chart-note or clearance letter from a primary care physician or hematologist 7. Significant psychiatric problems which might impair ability to give truly informed consent or which may impair follow-up communication with the surgeon and staff 8. Clinically significant cardiac arrhythmias are exclusionary unless there is a written clearance chart-note or clearance letter from a cardiologist 9. Heart/liver/kidney disease, neuropsychiatric disease classifying patient as ≥ ASA V 10. Major concomitant infections such as pneumonia or sepsis 11. In non-emergency surgery, pre-existing active bacterial skin infection at the time of the surgical incision; however, pre-existing bacterial infections are not exclusionary in burn or trauma patients.

12. Foreign material in the incision that cannot be removed 13. Recent systemic antimicrobial therapy 14. Clinically significant renal impairment or a creatinine clearance < 30 mL/min.

Vulnerable Subjects are excluded

1. Pregnant women
2. Nursing home residents, or other institutionalized persons are not fully alert, not cognizant or and not able to give informed consent are not eligible to participate as a research subject
3. Children < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of surgical site infections | 30 days

SECONDARY OUTCOMES:
Number of post-operative venous thromboembolism | 30 days
Amount of postoperative narcotic required | 7 days
Hospital length of stay | 30 days
Number of participants with adverse events | 24 hours